CLINICAL TRIAL: NCT00373347
Title: Identification of New Serum Diagnostic Markers of Hepatocellular Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-10767
Record Dates: First submitted 2006-09-06; First posted 2006-09-08 (Estimated); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to identify blood markers that have the ability to diagnose liver cancer with improved accuracy, so that it can be used alone or in conjunction with alpha-feto protein (AFP)

DETAILED DESCRIPTION:
Liver cancer is a deadly cancer that is typically hard to diagnose and treat. The currently used blood marker for the clinical diagnosis of liver cancer is alpha-feto protein (AFP), which misses 40-60% of patients with liver cancer because it lacks sufficient specificity and sensitivity. The purpose of this study is to identify blood markers that have the ability to diagnose liver cancer with improved accuracy, so that it can be used alone or in conjunction with AFP. The aim of this study is to identify new blood markers of liver cancer that can be used to increase the rate of accurate diagnosis of this malignancy.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with liver cancer based on biopsy or serum AFP level, associated with characteristic hypervascular liver tumors on triphasic spiral CT scan or MRI.
* Patients with non-cancer liver conditions such as cirrhosis, adenoma, cholangioma, or nodular hyperplasia.
* Patients with hepatitis B or hepatitis C viral infections not associated with liver cancer.

Exclusion Criteria:

-Patients will be excluded if, upon looking through their medical records, information required for data analysis are missing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with liver cancer
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2004-11; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Identify new blood markers of liver cancer | upto 12 months
  Blood specimens collected through another protocol, Patients would have signed informed consent for that protocol, and agreed to have their blood specimens stored for future research such as this one.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel So, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States